CLINICAL TRIAL: NCT00338819
Title: ActiveCare+SFT Hemodynamic Profile Compare to SCD Express in Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC06SP156CTIL
Record Dates: First submitted 2006-06-18; First posted 2006-06-20 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: DVT Prevention; Ventilated Patients
Keywords: DVT prevention; Hemodynamic study; IPC; CECT

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Purpose:

To test the hemodynamic profile generated by the MCS's ActiveCare+SFT device in ventilated patients and compare it to that of the Kendall SCD Express.

Design:

Comparative, prospective study. Patients are their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult ventilated patient (Age >18).
* The patient or his guardian is able and voluntarily prepared to sign the Informed Consent Form.

Exclusion Criteria:

* Known, preexisting DVT or PE.
* Patient who is participating in another clinical trial.
* Patient with contraindication to use of the device including patients with leg gangrene, recent skin graft or medical situations where increase venous and lymphatic return is undesirable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sorkine, Prof, Principal Investigator — Tel-Aviv Sourasky Medical Center